CLINICAL TRIAL: NCT02471534
Title: Study on Prediction of Fluid Responsiveness Using an Abdominal Compression-induced Change of Blood Pressure in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associated professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1411-061-6254
Record Dates: First submitted 2015-06-06; First posted 2015-06-15 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric patients with hypovolemia (Experimental): Right upper abdominal compression is performed in patients with hypovolemic signs including hypotension, decreased urine output and central venous pressure less than 5 mmHg. Changes of blood pressure during abdominal compression is continuously recorded.
  Interventions: Procedure: abdominal compression

INTERVENTIONS:
Procedure: abdominal compression — When there are clinical signs of hypovolemia, such as hypotension, decreased urine output and central venous pressure less than 5 mmHg, right upper abdomen is gently compressed for 10 seconds. Changes of blood pressure are continuously recorded during this period. About 3 min later, intravenous colloid fluid 10 mL/kg is infused for 20 min.

SUMMARY:
The purpose of this study is to evaluate predictability of an abdominal compression-induced change of blood pressure for fluid responsiveness in children.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate predictability of an abdominal compression-induced change of blood pressure for fluid responsiveness in children.

When there are clinical signs of hypovolemia, such as hypotension, decreased urine output and central venous pressure less than 5 mmHg, right upper abdomen is gently compressed for 10 seconds. Changes of blood pressure are continuously recorded during this period. About 3 min later, intravenous colloid fluid 10 mL/kg is infused for 20 min.

To evaluate the change of cardiac output, transesophageal or transthoracic echocardiography is performed before and after fluid administration. In addition, hemodynamic parameters including pulse pressure variation, systolic pressure variation, pleth variability index and central venous pressure are also recorded before and after fluid administration.

Finally, patients will be divided into fluid responder group and non-responder group. If cardiac output measured using echocardiography increases over 15% after fluid administration, the patient is fluid responder. Using ROC curve, diagnostic power of abdominal compression-induced blood pressure change for fluid responsiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing elective surgery, who require invasive blood pressure and central venous pressure monitoring during surgery

Exclusion Criteria:

* renal, hepatic and pulmonary disease
* preoperative infection: increased CPR, WBC over 10,000, and with fever
* genetic and hematologic disease
* intracardiac and extracardiac shunt
* single ventricle
* right heart dysfunction
* any intracardiac valve pathology
* increased intracranial pressure

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in cardiac index after volume expansion | before and after fluid administration (20 min)

SECONDARY OUTCOMES:
Changes in pleth variability index after volume expansion | before and after fluid administration (20 min)
Changes in respiratory changes of peak aortic blood flow velocities after volume expansion | before and after fluid administration (20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea